CLINICAL TRIAL: NCT04626934
Title: Can Specific Cognitive Intervention With Post-Acute Cognitively Impaired Hip Fracture Patients Improve Rehabilitation Outcome
Brief Title: Cognitive Intervention and Rehabilitation Outcomes in Hip Fracture Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, AVITAL HERSHKOVITZ, Head, Geriatric Rehabilitation Ward, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0465-20-RMC
Record Dates: First submitted 2020-10-22; First posted 2020-11-13 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hip Fracture; Rehabilitation; Cognitive Intervention
Keywords: cognitive; Intervention; Hip fracture; Rehabilitation; outcomes
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Randomized double blinded study
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the team that assess the patients do not know to which group the patients have been assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Patients in the control group will recieve conventional occupational therapy treatment: 3 weeks of all together 12 sessions, 45 minutes each.
  Interventions: Other: conventional occupational therapy treatment
- Intervention group (Experimental): The intervention will include all together 12 sessions, each being 45 minutes, for a total of 3 weeks. The intervention will include: 4 treatments in the area of memory and attention, 4 treatments in the area of problem solving, 4 treatments in the area of planning and analysing.
  Interventions: Other: specific cognitive intervention

INTERVENTIONS:
Other: specific cognitive intervention — The intervention will include all together 12 sessions, each being 45 minutes, for a total of 3 weeks. The intervention will include: 4 treatments in the area of memory and attention, 4 treatments in the area of problem solving, 4 treatments in the area of planning and analysing.
  Arms: Intervention group
Other: conventional occupational therapy treatment — The intervention will include all together 12 sessions of conventional occupational therapy treatments, each being 45 minutes, for a total of 3 weeks.
  Arms: control group

SUMMARY:
The objective of the present study is to assess whether specific cognitive intervention will influence rehabilitation outcomes of post-acute hip fracture patients.

DETAILED DESCRIPTION:
Hip fracture often occurs in frail older people and is a major concern for the health care systems because it is associated with an up to 36% excess mortality within 1 year. Hip fracture also represents a risk factor for further falls and fractures, functional decline and institutionalization, with <40% of hip fractured patients regaining their pre-injury level of ambulation.

One of the most challenging tasks of today's post-acute geriatric rehabilitation wards is improving the functional abilities of fragile hip-fractured patients and discharging most of them to their homes. Yet, the rising incidence of hip fractures in the elderly has created an overwhelming workload on those departments and has significantly increased the burden on healthcare resources. Previous studies have found that cognitive decline is an important negative predictor in rehabilitation. Several studies have shown that cognitive interventions can improve functional abilities of older people. Yet, these studies were conducted in community dwelling older people. Our study will assess this issue amongst post-acute rehabilitation hip fracture patients. Our hypotyhesis is that those patients recieving specific cognitive intervention will show significantly better rehabilitation outcomes and cognitive function.

The objective of the present study is to assess whether specific cognitive intervention will influence rehabilitation outcomes of post-acute hip fracture patients.

This is a randomized double blinded study. We will compare two groups: one will recieve specific cognitive intervention and a control group will recieve conventional occupational therapy treatment. Both groups will recieve the same amount of interventions.The interventions will include all together 12 sessions, each being 45 minutes, for a total of 3 weeks. The intervention will include: 4 treatments in the area of memory and attention, 4 treatments in the area of problem solving, 4 treatments in the area of planning and analysing.

Patients in the control group will recieve conventional occupational therapy treatment: 3 weeks of all together 12 sessions, 45 minutes each.

The outcome measures are: a disability measure, the Functional Independence Measure (FIM), the motor FIM, the Montebello Rehabilitation Factor Score (MRFS), also called motor FIM effectiveness. In addition 4 cognitive functional measures: the Color Trail Test, the Kettle Test, the Groningen Activity Restriction Skill (GARS), the Montreal Cognitive Assessment (MOCA).

The randomization process will be carried out by withdrawing a piece of paper written either A (intervention) (n=10) or B (control) (n=10) from an envelope. The subjects will not be informed as to which group they will be assigned. Patient recruitment and the randomization process will be supervised by the clinical staff. The assessors will be blinded to the type of intervention.

Statistical analysis will be performed using the IBM SPSS Statistics for Windows (Version 25.0. Armonk, NY: IBM Corp.).

The study sample size was estimated using the mean and the standard deviation of the motor FIM measure (calculated for this population), with improvement assumption by 7 points, with power of 0.8 and significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All concecutive hip fracture patients admitted to a post-acute rehabilitation ward Mini mental state examination above 17 Lived at home before the fracture and did not recieved 24 hour home aid

Exclusion Criteria:

* Patients who will not complete rehabilitation program due to worsening of their medical condition or unexpectedly cease rehabilitation will be omitted from the statistical analyses.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | The change in the measure from randomization until the date of discharge, assessed up 3 months.
  The FIM is a disability measure, administered on admission and upon discharge to assess change in functional abilities. The FIM comprises 18 parameters, each rated on a scale of 1 to 7 according to the degree of assistance required to perform a specific activity in 3 domains: activities of daily living (ADL) (8 parameters), mobility level (5 parameters) and cognitive function (5 parameters). The maximal total score for the FIM is 126. The patient's FIM score will be assessed during multi-disciplinary team meeting
motor Functional Independence Measure (mFIM) | The change in the measure from randomization until the date of discharge, assessed up 3 months.
  The motor FIM (mFIM) includes 13 parameters of ADL and mobility. maximal total score for the mFIM is 91. The patient's motor FIM score was assessed during multi-disciplinary team meeting
The Montebello Rehabilitation Factor Score (MRFS) | The score will be calculated at discharge, assessed up to 3 months from randomization.
  The MRFS achieved on the mFIM score is calculated by the Montebello Rehabilitation Factor Score (MRFS), designed to overcome the floor and ceiling effect problem and calculate each patient's specific potential for improvement. The MRFS also known as mFIM effectiveness, will be calculated as the mFIM score change (discharge mFIM score-admission mFIM score) divided by the mFIM maximum score (91) minus the mFIM admission score.

SECONDARY OUTCOMES:
Color Trail Test | The change in the measure from admission and upon completion of the intervention protocol (3 weeks).
  Assesses attention and visual perception and flexible thinking
Kettle Test | The change in the measure from admission and upon completion of the intervention protocol (3 weeks).
  Assesses working memory, attention, problem solving, praxis and safety
Groningen Activity Restriction Scale | The change in the measure from admission and upon completion of the intervention protocol (3 weeks).
  Assesses level of disability. This tool is comrised of 18 parameters each rated on a scale of 1 to 5. A low score shows higher functional level
Montreal Cognitive Assessement (MOCA) | The change in the measure from admission and upon completion of the intervention protocol (3 weeks).
  Assesses basic and executive cognitive skills. This tool includes 5 points related to executive function, 3 points to naming, 6 points to attention, 3 points to language use, 2 points to abstract thinking, 5 points to short term memory and 6 points to orientation. A score of 26 points and above shows normal cognitive functioning.
EQ-5D (EuroQol Group) | The change in the measure from admission and upon completion of the intervention protocol (3 weeks).
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. It ia applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys. EQ-5D is designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics, and in face-to-face interviews. It is cognitively undemanding, taking only a few minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Avital Hershkovitz, MD, Principal Investigator — Rabin MC
Locations (1):
- "Beit- Rivka" geriatric rehabilitation hospital, Petach Tiqva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adam S, Godlwana L, Maleka D. Changes in short-term cognitive function following a hip fracture in the elderly and the effect of cognitive function on early post-operative function. SA Orthopaedic Journal 2016;15:77-82.
- [Background] Oughli HA, Chen G, Philip Miller J, Nicol G, Butters MA, Avidan M, Stark S, Lenze EJ. Cognitive Improvement in Older Adults in the Year After Hip Fracture: Implications for Brain Resilience in Advanced Aging. Am J Geriatr Psychiatry. 2018 Nov;26(11):1119-1127. doi: 10.1016/j.jagp.2018.07.001. PMID 30454790
- [Background] Beloosesky Y, Grinblat J, Epelboym B, Weiss A, Grosman B, Hendel D. Functional gain of hip fracture patients in different cognitive and functional groups. Clin Rehabil. 2002 May;16(3):321-8. doi: 10.1191/0269215502cr497oa. PMID 12017519
- [Background] Rolland Y, Pillard F, Lauwers-Cances V, Busquere F, Vellas B, Lafont C. Rehabilitation outcome of elderly patients with hip fracture and cognitive impairment. Disabil Rehabil. 2004 Apr 8;26(7):425-31. doi: 10.1080/09638280410001663148. PMID 15204479
- [Background] Gruber-Baldini AL, Hosseini M, Orwig D, Grattan L, Chiles Shaffer N, Hochberg M, Magaziner J. Cognitive Differences between Men and Women who Fracture their Hip and Impact on Six-Month Survival. J Am Geriatr Soc. 2017 Mar;65(3):e64-e69. doi: 10.1111/jgs.14674. Epub 2017 Feb 8. PMID 28176306
- [Background] Mizrahi EH, Harel N, Heymann AD, Lubart E, Leibovitz A, Malik Gadot E, Barkan RB. The relation between gain in cognition during rehabilitation on functional outcome among hip fracture adult patients with and without pre- hip fracture dementia. Arch Gerontol Geriatr. 2018 Sep-Oct;78:177-180. doi: 10.1016/j.archger.2018.06.016. Epub 2018 Jun 30. PMID 30006209
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Lipardo DS, Tsang WW. Effects of combined physical and cognitive training on fall prevention and risk reduction in older persons with mild cognitive impairment: a randomized controlled study. Clin Rehabil. 2020 Jun;34(6):773-782. doi: 10.1177/0269215520918352. Epub 2020 May 7. PMID 32380917
- [Background] Lipardo DS, Tsang WWN. Falls prevention through physical and cognitive training (falls PACT) in older adults with mild cognitive impairment: a randomized controlled trial protocol. BMC Geriatr. 2018 Aug 24;18(1):193. doi: 10.1186/s12877-018-0868-2. PMID 30143002
- [Background] Reijnders J, van Heugten C, van Boxtel M. Cognitive interventions in healthy older adults and people with mild cognitive impairment: a systematic review. Ageing Res Rev. 2013 Jan;12(1):263-75. doi: 10.1016/j.arr.2012.07.003. Epub 2012 Jul 25. PMID 22841936
- [Background] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Background] Heruti RJ, Lusky A, Barell V, Ohry A, Adunsky A. Cognitive status at admission: does it affect the rehabilitation outcome of elderly patients with hip fracture? Arch Phys Med Rehabil. 1999 Apr;80(4):432-6. doi: 10.1016/s0003-9993(99)90281-2. PMID 10206606
- [Background] Hamilton BB, Granger CV, Sherwin FS, et al. A uniform national data system for medical rehabilitation. In: Fuhrer MJ, editor. Rehabilitation outcomes: analysis and measurement. Baltimore: Paul H Brooks Publishing Co; 1987. p 137-47.
- [Background] Granger CV, Hamilton BB. The Uniform Data System for Medical Rehabilitation report of first admissions for 1992. Am J Phys Med Rehabil. 1994 Feb;73(1):51-5. No abstract available. PMID 8305182
- [Background] Hartman-Maeir A, Erez AB, Ratzon N, Mattatia T, Weiss P. The validity of the Color Trail Test in the pre-driver assessment of individuals with acquired brain injury. Brain Inj. 2008 Dec;22(13-14):994-8. doi: 10.1080/02699050802491305. PMID 19117177
- [Background] Messinis L, Malegiannaki AC, Christodoulou T, Panagiotopoulos V, Papathanasopoulos P. Color Trails Test: normative data and criterion validity for the greek adult population. Arch Clin Neuropsychol. 2011 Jun;26(4):322-30. doi: 10.1093/arclin/acr027. Epub 2011 May 9. PMID 21558283
- [Background] Hartman-Maeir A, Harel H, Katz N. Kettle test--a brief measure of cognitive functional performance. Reliability and valdity in stroke rehabilitation. Am J Occup Ther. 2009 Sep-Oct;63(5):592-9. doi: 10.5014/ajot.63.5.592. PMID 19785258
- [Background] Harper KJ, Llewellyn K, Jacques A, Ingram K, Pearson S, Barton A. Kettle test efficacy in predicting cognitive and functional outcomes in geriatric rehabilitation. Aust Occup Ther J. 2019 Apr;66(2):219-226. doi: 10.1111/1440-1630.12540. Epub 2018 Oct 9. PMID 30298936
- [Background] Giambelluca E, Panigazzi M, Saade A, Imbriani M. Assessment of functional status and rehabilitative strategies in occupational therapy: role of the Groningen Activity Restriction Questionnaire. G Ital Med Lav Ergon. 2019 Mar;41(1):52-57. PMID 30946549
- [Background] Kempen GI, Miedema I, Ormel J, Molenaar W. The assessment of disability with the Groningen Activity Restriction Scale. Conceptual framework and psychometric properties. Soc Sci Med. 1996 Dec;43(11):1601-10. doi: 10.1016/s0277-9536(96)00057-3. PMID 8961404
- [Background] Markwick A, Zamboni G, de Jager CA. Profiles of cognitive subtest impairment in the Montreal Cognitive Assessment (MoCA) in a research cohort with normal Mini-Mental State Examination (MMSE) scores. J Clin Exp Neuropsychol. 2012;34(7):750-7. doi: 10.1080/13803395.2012.672966. Epub 2012 Apr 3. PMID 22468719
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759